CLINICAL TRIAL: NCT01044758
Title: Bridging Cognitive Aging in Rodents to Man Using fMRI in Amnestic MCI
Brief Title: Levetiracetam and Memory Function in Amnestic Mild Cognitive Impairment (MCI)
Status: Completed | Phase: Phase 2 | Type: Interventional
Sponsor: Johns Hopkins University (Other)
Collaborators: National Institute on Aging (NIA) (NIH)
Responsible Party: Sponsor
Allocation: Randomized | Model: Crossover | Masking: Double | Purpose: Basic Science
Other Study IDs: NA_00030573; RC2AG036419 (NIH)
Record Dates: First submitted 2010-01-07; First posted 2010-01-08 (Estimated); Results first posted 2017-08-21 (Actual); Last update posted 2017-08-21 (Actual); Status verified 2017-07

CONDITIONS: Mild Cognitive Impairment (MCI)
Keywords: Mild Cognitive Impairment; Amnestic Mild Cognitive Impairment; Functional Magnetic Resonance Imaging; Levetiracetam; Keppra; Medial Temporal Lobe; Memory Impairment; Alzheimer's Disease; AD
MeSH Terms: conditions — Cognitive Dysfunction; Memory Disorders; Alzheimer Disease | interventions — Levetiracetam

STUDY DESIGN:
Who Masked: Participant, Investigator
Oversight: Data Monitoring Committee: Yes

ARMS (7):
- aMCI_62.5mg drug first, then placebo (Experimental): Amnestic MCI:
  62.5mg levetiracetam twice daily (two weeks), washout (4 weeks), and placebo capsule twice daily (two weeks)
  Interventions: Drug: Levetiracetam 62.5mg; Drug: Placebo
- aMCI_Placebo first, then 62.5mg drug (Experimental): Amnestic MCI:
  Placebo capsule twice daily (two weeks), washout (4 weeks), and 62.5mg levetiracetam twice daily (two weeks)
  Interventions: Drug: Levetiracetam 62.5mg; Drug: Placebo
- aMCI_125mg drug first, then placebo (Experimental): Amnestic MCI:
  125mg levetiracetam twice daily (two weeks), washout (4 weeks), and placebo capsule twice daily (two weeks)
  Interventions: Drug: Levetiracetam 125mg; Drug: Placebo
- aMCI_Placebo first, then 125mg drug (Experimental): Amnestic MCI:
  Placebo capsule twice daily (two weeks), washout (4 weeks), and 125mg levetiracetam twice daily (two weeks)
  Interventions: Drug: Levetiracetam 125mg; Drug: Placebo
- aMCI_250mg drug first, then placebo (Experimental): Amnestic MCI: 250mg levetiracetam twice daily (two weeks), washout (4 weeks), and placebo capsule twice daily (two weeks)
  Interventions: Drug: Levetiracetam 250mg; Drug: Placebo
- aMCI_Placebo first, then 250mg drug (Experimental): Amnestic MCI:
  Placebo capsule twice daily (two weeks), washout (4 weeks), and 250mg levetiracetam twice daily (two weeks)
  Interventions: Drug: Levetiracetam 250mg; Drug: Placebo
- Control_Placebo first, then placebo (Placebo Comparator): Healthy control:
  placebo capsule twice daily (two weeks), washout (4 weeks), and placebo capsule twice daily (two weeks)
  Interventions: Drug: Placebo

INTERVENTIONS:
Drug: Levetiracetam 62.5mg — 62.5mg twice daily (2 weeks)
  Other Names: Keppra
  Arms: aMCI_62.5mg drug first, then placebo; aMCI_Placebo first, then 62.5mg drug
Drug: Levetiracetam 125mg — 125mg twice daily (2 weeks)
  Other Names: Keppra
  Arms: aMCI_125mg drug first, then placebo; aMCI_Placebo first, then 125mg drug
Drug: Levetiracetam 250mg — 250mg twice daily (2 weeks)
  Other Names: Keppra
  Arms: aMCI_250mg drug first, then placebo; aMCI_Placebo first, then 250mg drug
Drug: Placebo — placebo capsule twice daily (2 weeks)

SUMMARY:
This research is being done to find out if daily use of the drug levetiracetam can improve memory function in individuals with memory problems like those associated with Mild Cognitive Impairment (MCI) and Alzheimer's disease (AD).

DETAILED DESCRIPTION:
Increasing research is focused on conditions that precede the clinical diagnosis of Alzheimer's disease (AD) in order to detect patients at risk for early intervention. One such condition is mild cognitive impairment (MCI). Functional magnetic resonance imaging (fMRI) studies in this group of patients have reported increased activation in the Medial Temporal Lobe (MTL) during performance of memory tasks. The functional significance of increased activation is unclear. One possibility is that greater activity reflects the increased effort needed in order to maintain performance, and as such would be a compensatory response. An alternative possibility is that increased activation reflects aberrant physiology related to the disease process itself and as such would be a sign of greater underlying disease severity and would interfere with brain function.

Data in animal models suggest the possibility that low dose levetiracetam (well-tolerated anti-convulsant) treatment may reduce the observed hyperactivity and improve memory performance among individuals with MCI. The investigators are therefore conducting a within-subjects trial of 8 weeks duration, involving 144 subjects and low dose treatment with levetiracetam. During the course of the study, each subject may receive both drug and placebo for two weeks, with the order of administering those treatments counterbalanced. Cognitive testing and fMRI imaging will be obtained after 2-weeks on drug/placebo. The overall goal of the study is to determine if treatment of MCI subjects with low dose levetiracetam reduces hyperactivity within the MTL and improves memory performance.

ELIGIBILITY:
Inclusion Criteria:

* All: English as a first language; right handed; able to complete written informed consent.
* MCI subjects: In addition to above, must meet criteria for amnestic Mild Cognitive Impairment (MCI). This includes a memory complaint corroborated by an informant; impaired memory function for age and educational level; preserved general cognitive function; intact abilities of daily living; no clinical dementia.
* Age matched Controls: Must have memory and cognitive status that is normal for their age.

Exclusion Criteria:

* Familial Alzheimer's Disease (AD) due to known genetic mutations
* AD with Parkinsonian features; major psychiatric or behavioral disorders (e.g. depression, agitation, psychosis, manic-depressive disorder)
* Primary or metastatic intracranial neoplasm
* History of severe head trauma
* Intra-cerebral hemorrhage
* Seizure disorder
* Hemispheric stroke
* Presence of a progressive central nervous system disease
* Presence of lacunar infarcts
* Medical contraindications to MRI including cardiac pacemaker, presence of intraocular or intracranial metallic objects
* Any known allergy to levetiracetam or behavioral problems that are a contraindication to taking Levetiracetam (e.g. agitation)
* Prescribed use of anti-seizure medications.

Ages: 50 Years to 85 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 96 (Actual)
Dates: Start 2009-12; Primary Completion 2012-07 (Actual); Study Completion 2012-07 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Gregory L Krauss, MD, Principal Investigator — Johns Hopkins University
Locations (1):
- Johns Hopkins University School of Medicine, Baltimore, Maryland, United States

REFERENCES:
- [Background] Busche MA, Eichhoff G, Adelsberger H, Abramowski D, Wiederhold KH, Haass C, Staufenbiel M, Konnerth A, Garaschuk O. Clusters of hyperactive neurons near amyloid plaques in a mouse model of Alzheimer's disease. Science. 2008 Sep 19;321(5896):1686-9. doi: 10.1126/science.1162844. PMID 18802001
- [Background] Bakker A, Kirwan CB, Miller M, Stark CE. Pattern separation in the human hippocampal CA3 and dentate gyrus. Science. 2008 Mar 21;319(5870):1640-2. doi: 10.1126/science.1152882. PMID 18356518
- [Background] Palop JJ, Chin J, Roberson ED, Wang J, Thwin MT, Bien-Ly N, Yoo J, Ho KO, Yu GQ, Kreitzer A, Finkbeiner S, Noebels JL, Mucke L. Aberrant excitatory neuronal activity and compensatory remodeling of inhibitory hippocampal circuits in mouse models of Alzheimer's disease. Neuron. 2007 Sep 6;55(5):697-711. doi: 10.1016/j.neuron.2007.07.025. PMID 17785178
- [Background] Sperling R, Greve D, Dale A, Killiany R, Holmes J, Rosas HD, Cocchiarella A, Firth P, Rosen B, Lake S, Lange N, Routledge C, Albert M. Functional MRI detection of pharmacologically induced memory impairment. Proc Natl Acad Sci U S A. 2002 Jan 8;99(1):455-60. doi: 10.1073/pnas.012467899. Epub 2001 Dec 26. PMID 11756667
- [Background] Wilson IA, Ikonen S, Gallagher M, Eichenbaum H, Tanila H. Age-associated alterations of hippocampal place cells are subregion specific. J Neurosci. 2005 Jul 20;25(29):6877-86. doi: 10.1523/JNEUROSCI.1744-05.2005. PMID 16033897
- [Background] Wilson IA, Gallagher M, Eichenbaum H, Tanila H. Neurocognitive aging: prior memories hinder new hippocampal encoding. Trends Neurosci. 2006 Dec;29(12):662-70. doi: 10.1016/j.tins.2006.10.002. Epub 2006 Oct 13. PMID 17046075
- [Background] Koh MT, Haberman RP, Foti S, McCown TJ, Gallagher M. Treatment strategies targeting excess hippocampal activity benefit aged rats with cognitive impairment. Neuropsychopharmacology. 2010 Mar;35(4):1016-25. doi: 10.1038/npp.2009.207. Epub 2009 Dec 23. PMID 20032967

RESULTS

PARTICIPANT FLOW:
Pre-assignment Details: Data for the 125mg BID treatment cohort was collected first. Analysis showed no effects of treatment order. As a result, data was collapsed and analyzed irrespective of order across all doses. All subsequent data analyses are thus provided collapsed across treatment orders in all reporting on this study, including the results reported here.
Period: Overall Study
Arm/Group | aMCI_62.5mg Drug First, Then Placebo | aMCI_Placebo First, Then 62.5mg Drug | aMCI_125mg Drug First, Then Placebo | aMCI_Placebo First, Then 125mg Drug | aMCI_250mg Drug First, Then Placebo | aMCI_Placebo First, Then 250mg Drug | Control_Placebo First, Then Placebo
Started | 12 | 12 | 11 | 12 | 11 | 11 | 27
Completed | 8 | 12 | 7 | 10 | 9 | 8 | 17
Not Completed | 4 | 0 | 4 | 2 | 2 | 3 | 10

BASELINE CHARACTERISTICS:
Groups:
- Control_Placebo First, Then Placebo: Healthy control
  placebo capsule twice daily (two weeks), washout (4 weeks), and placebo capsule twice daily (two weeks)
- Total: Total of all reporting groups
Arm/Group | aMCI_62.5mg Drug First, Then Placebo | aMCI_Placebo First, Then 62.5mg Drug | aMCI_125mg Drug First, Then Placebo | aMCI_Placebo First, Then 125mg Drug | aMCI_250mg Drug First, Then Placebo | aMCI_Placebo First, Then 250mg Drug | Control_Placebo First, Then Placebo | Total
Number analyzed (Participants) | 8 | 12 | 7 | 10 | 9 | 8 | 17 | 71
Age, Categorical [Count of Participants; unit: Participants]
  <=18 years | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
  Between 18 and 65 years | 0 | 2 | 2 | 0 | 1 | 1 | 1 | 7
  >=65 years | 8 | 10 | 5 | 10 | 8 | 7 | 16 | 64
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 5 | 6 | 6 | 5 | 5 | 6 | 8 | 41
  Male | 3 | 6 | 1 | 5 | 4 | 2 | 9 | 30
Region of Enrollment [Number; unit: participants]
  United States | 8 | 12 | 7 | 10 | 9 | 8 | 17 | 71

OUTCOME MEASURES:

1. Primary Outcome: Brain Activity in the Dentate Gyrus / CA3 Subregion of the Hippocampus Measured With Blood Oxygenation Level Dependent (BOLD) Functional MRI
Description: Measurement of average brain activity in the dentate gyrus / CA3 subregion of the hippocampus measured with BOLD functional MRI in patients with mild cognitive impairment on placebo and on drug compared to average brain activity in this brain area in control subjects.
Time Frame: 2 weeks
Measure: Mean (Standard Error); unit: mean beta coefficient
Groups:
- aMCI_62.5: 62.5 mg levetiracetam twice daily for two weeks
- aMCI_62.5 Placebo: 62.5mg levetiracetam placebo comparator
- aMCI_125: 125 mg Levetiracetam twice daily for two weeks.
- aMCI_125 Placebo: 125mg levetiracetam placebo comparator
- aMCI_250: 250mg levetiracetam twice daily for two weeks
- aMCI_250 Placebo: 250mg levetiracetam placebo comparator
- Age Matched Control: Placebo capsule twice daily for two weeks
Arm/Group | aMCI_62.5 | aMCI_62.5 Placebo | aMCI_125 | aMCI_125 Placebo | aMCI_250 | aMCI_250 Placebo | Age Matched Control
Number analyzed (Participants) | 20 | 20 | 17 | 17 | 17 | 17 | 17
mean beta coefficient | -0.1203 (0.3475) | 0.4353 (0.2215) | -0.2238 (0.1747) | 0.8814 (0.3798) | 0.3928 (0.2366) | 0.4825 (0.1954) | -.02507 (.2238)

2. Secondary Outcome: Behavioral Performance as Assessed in the Functional Magnetic Resonance Imaging (fMRI) Memory Task
Description: Mnemonic similarity task which assesses long term memory function. Scale ranges from 0-100 with higher scores indicating better memory performance.
Time Frame: 2 weeks
Measure: Mean (Standard Error); unit: percent correct recalled
Groups:
- aMCI_62.5: 62.5mg levetiracetam twice daily for two weeks
- aMCI_62.5 Placebo: 62.6mg levetiracetam placebo comparator
- aMCI_125: 125mg levetiracetam twice daily for two weeks
Arm/Group | aMCI_62.5 | aMCI_62.5 Placebo | aMCI_125 | aMCI_125 Placebo | aMCI_250 | aMCI_250 Placebo | Age Matched Control
Number analyzed (Participants) | 20 | 20 | 17 | 17 | 17 | 17 | 17
percent correct recalled | 38 (4) | 33 (5) | 33 (5) | 28 (4) | 34 (4) | 31 (3) | 44 (4)

ADVERSE EVENTS:
Groups:
- aMCI_62.5 Placebo: 62.5 mg placebo comparator (placebo capsule twice daily for two weeks)
- aMCI_125 Placebo: 125 mg placebo comparator (placebo capsule twice daily for two weeks)
- aMCI_250: 250 mg levetiracetam twice daily for two weeks
- aMCI_250 Placebo: 250 mg placebo comparator (placebo capsule twice daily for two weeks)
Arm/Group | aMCI_62.5 | aMCI_62.5 Placebo | aMCI_125 | aMCI_125 Placebo | aMCI_250 | aMCI_250 Placebo | Age Matched Control
All-Cause Mortality (participants affected / at risk) | 0/24 | 0/24 | 0/23 | 0/23 | 0/22 | 0/22 | 0/27
Serious Adverse Events (participants affected / at risk) | 0/24 | 0/24 | 0/23 | 0/23 | 0/22 | 0/22 | 0/27
Other Adverse Events (participants affected / at risk) | 5/24 | 0/24 | 3/23 | 0/23 | 5/22 | 7/22 | 3/27
OTHER ADVERSE EVENTS (reported when occurring in more than 5% of participants in an arm); cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | aMCI_62.5 (N=24) | aMCI_62.5 Placebo (N=24) | aMCI_125 (N=23) | aMCI_125 Placebo (N=23) | aMCI_250 (N=22) | aMCI_250 Placebo (N=22) | Age Matched Control (N=27)
somnolence (Nervous system disorders) | 5 (7) | 0 (0) | 3 (3) | 0 (0) | 5 (6) | 4 (6) | 3 (3)
Irritability (General disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 3 (3) | 0 (0)

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: No